CLINICAL TRIAL: NCT05569031
Title: A Comparative Study of the Efficacy of Venlafaxine and Naltrexone for Relapse Prevention in Patients With Opioid Use Disorder Attributed to Tramadol
Brief Title: Treatment of Withdrawal Symptoms and Prevention of Relapse in Patients With Tramadol Abuse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Medhat Bassiony, Professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4853
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Opiate Withdrawal Syndrome
Keywords: tramadol abuse; withdrawal; lofixidine; venlaaxine
MeSH Terms: interventions — Venlafaxine Hydrochloride; lofexidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- venlafaxidine (Active Comparator): venlafaxine 75-225 mg per day.
  Interventions: Drug: Venlafaxine
- Lofixidine (Active Comparator): Lofixidine 1.6 to 2.4 per day.
  Interventions: Drug: Lofexidine

INTERVENTIONS:
Drug: Venlafaxine — patients with tramadol abuse will use venlafaxine for 10 days.
  Arms: venlafaxidine
Drug: Lofexidine — patients with tramadol abuse will use lofixidine for 10 days.
  Arms: Lofixidine

SUMMARY:
Tramadol abuse is a public health problem in Egypt. There are no approved medications for treatment of withdrawal symptoms or prevention of relapse in patients with tramadol abuse. The objective of this study was to compare the efficacy of venlafaxine and lofixidine in treating the withdrawal symptoms and to compare between venlafaxine and naltrexone in relapse prevention of tramadol abuse. Patients with tramadol abuse will be divided randomly to use venlafaxine or lofixidine after discontinuation of tramadol. The efficacy will be measured by the Clinical Opiate Withdrawal Scale. The medications will be used for 10 days after discontinuation of tramadol. After the detoxification stage, patients who used venlafaxine will continue to use it while patients who used lofixidine will use naltrexone during the relapse prevention phase (2 months).

DETAILED DESCRIPTION:
Introduction Venlafaxine is a nontricyclic antidepressant that selectively inhibits serotonin reuptake at low doses, but at higher doses, it blocks neuronal reuptake of serotonin, norepinephrine, and, to a lesser degree, dopamine (Debonnel et al., 2007).

Venlafaxine was also proved to have analgesic and antinociceptive effects through opioid mechanisms (Markowitz & Patrick, 1998; Schreiber et al., 1999; Schreiber et al., 2002).

In the study of McDowell et al. (2000), venlafaxine was successfully used to treat patients with cocaine dependence comorbid with major depression. In animal studies, venlafaxine demonstrated effectiveness to attenuate morphine withdrawal symptoms (Lu et al., 2001) and attenuate acquisition of intravenous self-administration of heroin in rats (Magalas et al., 2005). Lin et al. (2008) found that venlafaxine is effective in alleviating withdrawal symptoms of heroin with good tolerability and safety.

Lofixidine works by blocking the release of norepinephrine, a hormone similar to adrenaline that contributes to opioid withdrawal symptoms. Lofexidine is a non-opioid prescription medicine used in adults to help with the symptoms of opioid withdrawal that may happen when you stop taking an opioid suddenly.

Naltrexone, is an opioid antagonist, without abuse liability and the oral formulation was found to be a safe option for motivated individuals who prefer not to be treated with opioid agonist medication or where opioid agonist medications are not legally available (Krupitsky et al., 2010, Ling et al., 2012, Mooney, 2016). Although oral naltrexone had a limited side effect profile, the clinical evidence demonstrating its efficacy for the treatment of opioid use disorder has revealed limitations in its use, particularly as it requires detoxification and a several days period of opioid abstinence prior to initiation (Ling et al., 2012, Nunes et al., 2015, Mooney, 2016).

Rational Tramadol abuse is a public health problem in Egypt affecting both adults and adolescents. Dissatisfaction with current available regimens for treatment of tramadol abuse has led to the search for alternatives. This study will investigate the efficacy and tolerability of venlafaxine versus lofexidine for management of withdrawal symptoms of tramadol abuse and venlafaxine versus naltrexone in preventing relapse.

Research question:

* Is venlafaxine as effective as lofexidine for treatment of tramadol withdrawal symptoms?
* Is venlafaxine as effective as naltrexone in relapse prevention of tramadol abuse?

HYPOTHESIS:

We assume that venlafaxine is as effective as lofexidine for treatment of tramadol withdrawal symptoms and as effective as naltrexone in prevention of tramadol relapse.

AIM:

- This study aims at finding an effective and safe treatment for patients with tramadol abuse.

OBJECTIVES:

1. To compare the efficacy of venlafaxine versus lofexidine for treatment of tramadol withdrawal symptoms.
2. To compare the efficacy of venlafaxine versus naltrexone in prevention of tramadol relapse.

SUBJECTS AND METHODS:

I -Technical design This study was be carried out at the outpatient clinics and inpatient wards of addiction unit at Zagazig university hospitals, Egypt.

Sample size Assuming that the mean number of opioid negative tests in a previous study comparing buprenorphine and naltrexone in relapse prevention was 19.7+_6.1 for buprenorphine VS 15.4+_4.9 for naltrexone. The sample was estimated to be 52 cases of tramadol abuse (26 cases in each treatment group) with 95% confidence interval and 80% test power (open epi program).

II-Operational design:

This was a a randomized comparative clinical trial, which included 52 patients with tramadol abuse who were divided randomly into 2 groups:

Detoxification stage (10 days) Group 1: patients received venlafaxine xr 75mg once daily + symptomatic treatment.

Group 2: received lofexidine .2mg ( 0.8 - 1.6 mg per day) + symptomatic treatment.

Relapse prevention stage (2 month) Group 1: patients continued to use venlafaxine xr, which increased gradually on weekly intervals to 225 mg/d Group 2: patients used naltrexone 50mg/d The diagnosis of tramadol abuse and any comorbid psychiatric disorder was based on the Structured Clinical Interview for DSM-IV axis I disorders (SCID-I) done on Day 1 of the study (First et al., 2012). The severity of withdrawal symptoms was assessed using the Clinical Opiate Withdrawal Scale (COWS) done on day 3 and 10 of the study (Wesson & Ling, 2003). Hamilton anxiety rating scale (HAM-A) (Hamilton, 1959), Hamilton depression rating scale (HAM-D) (Hamilton, 1960) and Beck Depression Inventory (Beck et al., 1996) were used to assess anxiety and depressive symptoms on day 1 and at the end of the study after 2 months. Urine screen for drugs of abuse was done twice weekly to verify abstinence. Craving was assessed monthly. Outcome measures were treating tramadol withdrawal symptoms, the retention rate in every group and the result of urine screen test at the end of the study.

III-Administrative design:

1. Approval was obtained from the Institutional Review Board (IRB) and the Department of Psychiatry, Zagazig University, Egypt.
2. A written consent was signed by the study participants.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. All patients should meet DSM-IV criteria for opioid use disorder.
2. Both genders will be included.
3. Age will be above 18 years.
4. All socioeconomic classes and educational levels will be included.

Exclusion criteria:

1. Age: 18 years or below.
2. Presence of mental retardation, dementia or delirium. .
3. Pregnancy or lactation.
4. Known history of allergy, adverse effects or sensitivity to the study medication.
5. Unstable psychiatric or medical condition.
6. Immediate suicide risk.
7. Regular use of psychoactive drugs or dependence on substances other than opioids, nicotine, or caffeine.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
detoxification stage | 10 days
  the efficacy was measured by decrease in the score of the "Clinical Opiate Withdrawal Scale (COWS). Increase in the score means worsening and score decrease means improvement. We compared the mean + SD for all groups. COWS Score: 5- 12 = mild; 1 3-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal.

SECONDARY OUTCOMES:
Relapse prevention | 2 months
  This outcome was measured by the number of patients who remains in treatment and have negative urine screen for tramadol.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bassiony MM, Abdelfattah NR, Elshabrawy A, Adly MM. A comparative study of the efficacy of venlafaxine and naltrexone for relapse prevention in patients with opioid use disorder attributed to tramadol. Int Clin Psychopharmacol. 2024 Nov 1;39(6):341-349. doi: 10.1097/YIC.0000000000000487. Epub 2023 Sep 20. PMID 37729663